CLINICAL TRIAL: NCT05683938
Title: GentleCath™ Air Intermittent Catheter Smartwatch Real Life Pilot Study
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-19-400
Record Dates: First submitted 2022-07-22; First posted 2023-01-13 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Neurogenic Bladder
Keywords: neurogenic bladder; intermittent self-catherterisation
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intermittent self-catheterisation — GentleCath™ Air intermittent catheter

SUMMARY:
As part of the ongoing Clinical Evaluation and Post Market Clinical Follow Up (PMCF) activities it was determined that a pilot study should be conducted to look at how real life data such as various physiological measurements can be collected via a Smart-Watch during intermittent self-catheterisation whilst also collecting real life feedback from users on comfort as measured by levels of possible discomfort and on levels of anxiety which may be associated with intermittent catheterisation over a period of time.

Adherence to catheter regimen and proper emptying of the bladder is of clinical relevance for clean intermittent catheterisation. A Daily Fluid Diary is included in this pilot study together with the use of the microphone of the Apple™ Smart Watch to investigate the feasibility of tracking input and output of fluids. The user acceptance of the Daily Fluid Diary offered via the iPhone app and the feasibility of the microphone to capture bladder emptying or voiding are to be tested within this pilot.

ELIGIBILITY:
Inclusion Criteria:

* • Females aged 18 years old and above who require intermittent bladder drainage

  * Idiopathic and Neurogenic subjects
  * Be willing and able to provide electronic informed consent
  * Be willing and able to wear a Polar H10 chest-strap
  * Must be willing and able to use the smart technology provided e.g. Smart Phone with software application and/or smart watch to answer the required questions
  * Currently use intermittent catheters
  * Have used intermittent catheters for more than 6 months
  * Subjects who perform intermittent catheterisation at least twice per day
  * Speak, read and write in English

Exclusion Criteria:

* • Subjects who require intermittent catheterisation to administer irrigation or instillation.

  * Short term voiding difficulties following Botox injections
  * Currently participating in another clinical trial or has participated in a clinical study in the previous month
  * Current users of the GentleCath™ Air intermittent catheter
  * Exhibiting any other medical condition which, according to the investigator, justifies the subject's exclusion from the study, for example- medical conditions that affect heart rate, anxiety disorders, uncontrolled diabetes, hyperthyroidism, psychological disorders, and other causes of blunted autonomic response.
  * Subjects with a known alcohol dependency and/or recreational drug use
  * Current symptomatic Urinary Tract Infection (UTI) or diagnosed UTI in the previous 2 weeks
  * Known sensitivity to the catheter device components or the Apple™ Watch or Polar™ H10 chest straps
  * Pregnancy or breast feeding
  * Subjects, in the opinion of the Investigator, unable to carry out the study procedures or other factors e.g. Planned surgery which may prevent them from completing the study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females (Idiopathic and Neurogenic) aged 18 years old and above who require intermittent bladder drainage
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
To collect physiological measurements associated with self-catheterisation using an Apple™ Watch 6.0, an iPhone SE 2020 and a Polar H10 chest-strap plus a software application | 28 days
  Measurements of Heart Rate (variability) will be collected using the Polar H10 chest strap

SECONDARY OUTCOMES:
To obtain user feedback, in a Real-Life setting, on the comfort as measured by the level of discomfort in the use of GentleCath™ Air intermittent catheter and related QoL and anxiety associated with self-catheterisation in general | 28 days
  A questionnaire geared towards comfort and quality of life will be completed with self-catheterization, changes in scores will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No